CLINICAL TRIAL: NCT04122391
Title: Patterns of Inattentional Blindness During Perioperative Cardiac Arrest: Do Healthcare Providers See and Correct Critical Errors?
Brief Title: Intentional Blindness During Perioperative Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KidSIM Simulation Program (Network)
Responsible Party: Sponsor
Other Study IDs: REB19-1549
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Arrest
Keywords: simulation; cardiac arrest; perioperative cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: team will work in OR with volume of 85 dB
  Interventions: Other: sound level volume
- intervention: team will work in OR with volume of 100 dB
  Interventions: Other: sound level volume

INTERVENTIONS:
Other: sound level volume — Noise level during cardiac arrest

SUMMARY:
Cardiac arrest in the operating room is a rare but potentially catastrophic event with mortality rates greater than 50%. Recent CPR guidelines published by the American Heart Association (AHA) and the Heart and Stroke Foundation of Canada (HSFC) describe how high quality CPR improves survival rates and neurological outcomes from cardiac arrest. Despite CPR training, adherence rates with performance guidelines are alarmingly low in many pediatric hospitals . In addition to performance errors, medication errors have been reported to be as high as 50% during cardiopulmonary arrest. This can be attributed to many factors, including distractions and poor communication among team members. Previous studies suggested that loud noise in the operating room caused poor communication and impaired surgical performance. To understand more about simulation awareness during peri-operative cardiac arrest, the investigators are planning on conducting a prospective observational study, using a simulated perioperative cardiac arrest scenario in pediatric hospital.The investigators are aiming for a convenient sample of 20 simulation sessions. Each session will have a team of CPR providers (2 participants and 4 confederates). The 2 participants will include one anesthesiologist and one operating room nurse. The participants will be randomized into two group; group A will work in a noise environment of 85 dBA ( as per recommendation by the National Institute for Occupational Safety and Health (NIOSH), and group B will work in a noise environment of 100 dBA. Participants will be wearing eye tracking devices during the scenario (Tobii Pro GlassesTM) designed to capture areas of interest (AOI) / visual fixation. The investigators hypothesize that CC and medication errors are frequently left undetected and uncorrected, and that the less noise distractions during resuscitation improves but does not eliminate this pattern of inattentional blindness in resuscitation teams during simulated perioperative pediatric cardiac arrest. They also hypothesize that "look but not act" events are a frequent occurrence during simulated pediatric cardiac arrest, and that healthcare providers will have varying reasons that explain the occurrence of "look but not act" events.

DETAILED DESCRIPTION:
Pediatric Cardiac Arrest and intraoperative arrest Cardiac arrest in the operating room is a rare but potentially catastrophic event with mortality rate of more than 50% . Each year, it is estimated that >15,000 infants and children in North America receive cardiopulmonary resuscitation (CPR) as a treatment of cardiopulmonary arrest (CPA). The incidence of pediatric perioperative cardiac arrest can be as high as 20.9 per 10,000 cases. Recent CPR guidelines published by the American Heart Association (AHA) and the Heart and Stroke Foundation of Canada (HSFC) describe how high quality chest compressions (CC) with adequate compression depth (5-6 cm) and rate (100-120 beats/min) improves survival rates and neurological outcomes from CPA. Patients receiving CC with adequate depth are more likely to survive than those who aren't (70% vs 16% 24-hour survival), while those receiving CC within the target rate range demonstrate the highest rates of survival.

Despite CPR training, adherence rates with performance guidelines are alarmingly low at pediatric hospitals. Professional rescuers observed that CPR quality during simulated and real cardiac arrests frequently fall well short of guidelines in leading institutions. In addition to performance errors, medication errors have been reported to be as high as 50% during cardiopulmonary arrest. Because of the resuscitation environment, errors in prescribing, doing, preparing, labeling and administering the drugs are prone to occur. A 2015 Institute of Medicine (IOM) Report entitled: "Strategies to Improve Cardiac Arrest Survival: A Time to Act", recommended translational research focusing on the function of resuscitation teams be undertaken to improve outcomes from CPA.

1) Goals, Objectives, and Project Outputs Goal To identify, describe and quantify patterns of inattentional blindness related to critical errors for resuscitation teams during the management of perioperative pediatric cardiac arrest.

Objectives

1. To determine the frequency of CC-related errors that are undetected by resuscitation teams during management of a simulated pediatric cardiac arrest with average noise level (85 dBA) vs high noise (100 dBA) in the operating room during resuscitation.
2. To determine the frequency of medication-related errors that are undetected by resuscitation teams during management of a simulated pediatric cardiac arrest with average noise level (85dBA) vs high noise (100 dBA) level in the operating room during resuscitation.
3. To determine the frequency of "look but not act" events (for CC related errors/ medication) during the management of simulated perioperative cardiac arrest.
4. To describe the underlying cause for "look but not act" events as it relates to CC related errors in management of simulated perioperative cardiac arrest.

Proposed Project Outputs

1. The investigators hypothesize that CC and medication errors are frequently left undetected and uncorrected, and that the less noise distractions during resuscitation improves but does not eliminate this pattern of inattentional blindness in resuscitation teams during simulated perioperative pediatric cardiac arrest.
2. They hypothesize that "look but not act" events are a frequent occurrence during simulated pediatric cardiac arrest, and that healthcare providers will have varying reasons that explain the occurrence of "look but not act" events.

ELIGIBILITY:
Inclusion Criteria:

1. current PALS certification or PALS instructor
2. attending physician or senior resident (year 3 or 4) or fellow in pediatric anesthesia.
3. The other provider will be OR nurse with recent basic life support certification (past 1 year).

Exclusion Criteria:

* participant refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anesthesia (Staff, fellows, senior residents) OR nursing staff
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
proportion of each error type detected by any participant member of the resuscitation team (ie. team leader, the OR nurse). | simulation time = 10 minutes
  Detection is defined as one or more participant member of the resuscitation team either: (a) verbally stating and sharing nature of error with one or more team members (eg. "the CC rate seems slow"); and/or (b) verbally providing corrective feedback for the specific error (eg. "Please press faster to improve CC rate").

SECONDARY OUTCOMES:
Time spent to detect the error | 30 seconds
  time for the participant to detect international errors
Team lead fixation errors | 1 minute
  Duration and number of visual fixations on pre-defined areas of interest (AOI) for each error type by team leader and team members, as measured by eye tracking devices
Frequency of "look but not act" | 45 minutes
  Frequency of "look but not act" events for each error type - the participant(s) looks at the AOI for the error, but does not act (as determined by video review)
Reasons for "look but not act | 45 minutes
  Reasons for "look but not act" events will be captured during semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Cheng, Study Director — University of Calgary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gonzalez LP, Braz JR, Modolo MP, de Carvalho LR, Modolo NS, Braz LG. Pediatric perioperative cardiac arrest and mortality: a study from a tertiary teaching hospital. Pediatr Crit Care Med. 2014 Nov;15(9):878-84. doi: 10.1097/PCC.0000000000000248. PMID 25226499
- [Background] de Caen AR, Berg MD, Chameides L, Gooden CK, Hickey RW, Scott HF, Sutton RM, Tijssen JA, Topjian A, van der Jagt EW, Schexnayder SM, Samson RA. Part 12: Pediatric Advanced Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S526-42. doi: 10.1161/CIR.0000000000000266. No abstract available. PMID 26473000
- [Background] de Caen AR, Maconochie IK, Aickin R, Atkins DL, Biarent D, Guerguerian AM, Kleinman ME, Kloeck DA, Meaney PA, Nadkarni VM, Ng KC, Nuthall G, Reis AG, Shimizu N, Tibballs J, Veliz Pintos R; Pediatric Basic Life Support and Pediatric Advanced Life Support Chapter Collaborators. Part 6: Pediatric Basic Life Support and Pediatric Advanced Life Support: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2015 Oct 20;132(16 Suppl 1):S177-203. doi: 10.1161/CIR.0000000000000275. No abstract available. PMID 26472853
- [Background] Meaney PA, Bobrow BJ, Mancini ME, Christenson J, de Caen AR, Bhanji F, Abella BS, Kleinman ME, Edelson DP, Berg RA, Aufderheide TP, Menon V, Leary M; CPR Quality Summit Investigators, the American Heart Association Emergency Cardiovascular Care Committee, and the Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation. Cardiopulmonary resuscitation quality: [corrected] improving cardiac resuscitation outcomes both inside and outside the hospital: a consensus statement from the American Heart Association. Circulation. 2013 Jul 23;128(4):417-35. doi: 10.1161/CIR.0b013e31829d8654. Epub 2013 Jun 25. PMID 23801105
- [Background] Hinkelbein J, Andres J, Thies KC, DE Robertis E. Perioperative cardiac arrest in the operating room environment: a review of the literature. Minerva Anestesiol. 2017 Nov;83(11):1190-1198. doi: 10.23736/S0375-9393.17.11802-X. Epub 2017 Mar 28. PMID 28358179
- [Background] Sutton RM, French B, Niles DE, Donoghue A, Topjian AA, Nishisaki A, Leffelman J, Wolfe H, Berg RA, Nadkarni VM, Meaney PA. 2010 American Heart Association recommended compression depths during pediatric in-hospital resuscitations are associated with survival. Resuscitation. 2014 Sep;85(9):1179-84. doi: 10.1016/j.resuscitation.2014.05.007. Epub 2014 May 16. PMID 24842846
- [Background] Idris AH, Guffey D, Aufderheide TP, Brown S, Morrison LJ, Nichols P, Powell J, Daya M, Bigham BL, Atkins DL, Berg R, Davis D, Stiell I, Sopko G, Nichol G; Resuscitation Outcomes Consortium (ROC) Investigators. Relationship between chest compression rates and outcomes from cardiac arrest. Circulation. 2012 Jun 19;125(24):3004-12. doi: 10.1161/CIRCULATIONAHA.111.059535. Epub 2012 May 23. PMID 22623717
- [Background] Idris AH, Guffey D, Pepe PE, Brown SP, Brooks SC, Callaway CW, Christenson J, Davis DP, Daya MR, Gray R, Kudenchuk PJ, Larsen J, Lin S, Menegazzi JJ, Sheehan K, Sopko G, Stiell I, Nichol G, Aufderheide TP; Resuscitation Outcomes Consortium Investigators. Chest compression rates and survival following out-of-hospital cardiac arrest. Crit Care Med. 2015 Apr;43(4):840-8. doi: 10.1097/CCM.0000000000000824. PMID 25565457
- [Background] Sutton RM, Maltese MR, Niles D, French B, Nishisaki A, Arbogast KB, Donoghue A, Berg RA, Helfaer MA, Nadkarni V. Quantitative analysis of chest compression interruptions during in-hospital resuscitation of older children and adolescents. Resuscitation. 2009 Nov;80(11):1259-63. doi: 10.1016/j.resuscitation.2009.08.009. Epub 2009 Sep 4. PMID 19733427
- [Background] Sutton RM, Niles D, French B, Maltese MR, Leffelman J, Eilevstjonn J, Wolfe H, Nishisaki A, Meaney PA, Berg RA, Nadkarni VM. First quantitative analysis of cardiopulmonary resuscitation quality during in-hospital cardiac arrests of young children. Resuscitation. 2014 Jan;85(1):70-4. doi: 10.1016/j.resuscitation.2013.08.014. Epub 2013 Aug 29. PMID 23994802
- [Background] Sutton RM, Niles D, Nysaether J, Abella BS, Arbogast KB, Nishisaki A, Maltese MR, Donoghue A, Bishnoi R, Helfaer MA, Myklebust H, Nadkarni V. Quantitative analysis of CPR quality during in-hospital resuscitation of older children and adolescents. Pediatrics. 2009 Aug;124(2):494-9. doi: 10.1542/peds.2008-1930. Epub 2009 Jul 5. PMID 19581266